CLINICAL TRIAL: NCT06862648
Title: Pivotal Study of the SUI-100™ for the Treatment of Stress Urinary Incontinence (SUI): A Nonsignificant Risk (NSR) Device (SaHARA) Study
Brief Title: Evaluating SUI-100™, A Non-Invasive Device for the Treatment of Stress Urinary Incontinence
Acronym: SaHARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acoustic Wave Cell Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SaHARA/SUI-003
Record Dates: First submitted 2025-02-12; First posted 2025-03-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: Stress Urinary Incontinence; Female Urinary Incontinence; Mild-to-Moderate SUI; Urine Leakage; Acoustic Energy Therapy; Non-Invasive Treatment; SUI-100 Device; Pivotal Study; Randomized Controlled Trial (RCT); Sham-Controlled Trial; Blinded Study; Multicenter Study; 24-Hour Pad Weight Test; Reduction in Urine Leakage; Improved Quality of Life; Symptom Improvement; Incontinence Impact Questionnaire (IIQ-7); Adverse Event Monitoring; Device Safety Evaluation; IRB Oversight; Female Participants; Ages 22-70; Non-Surgical Candidates; Conservative Treatment Options; Baseline Assessments; Treatment Phase; Follow-Up Phase; Maintenance Phase; Semi-Weekly Treatments; Crossover Option; Low-Risk Intervention
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Randomized with option for crossover: Participants assigned to the sham arm will have the option to crossover and receive active treatments after the unblinding phase.
Who Masked: Participant, Investigator
Masking Description: The principal investigator will remain blinded until study unblinding occurs. Study staff will assemble the machine before each session so that the participant will only see the device in the assembly for which they are assigned (active or sham).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Active Treatment Arm (Experimental): Participants receive active sessions using the SUI-100 Device.
  Interventions: Device: Acoustic Stimulation Therapy Device
- Sham Treatment Arm (Sham Comparator): Participants receive sham sessions using the SUI-100 Device.
  Interventions: Device: Sham Acoustic Stimulation Therapy Device
- Crossover Active Treatment Arm (Experimental): Sham participants who opt to crossover after unblinding receive active sessions with the SUI-100 Device.
  Interventions: Device: Acoustic Stimulation Therapy Device

INTERVENTIONS:
Device: Acoustic Stimulation Therapy Device — The SUI-100 Device is a non-invasive device designed for the treatment of stress urinary incontinence (SUI) in females.
  Other Names: SUI-100™ Device
  Arms: Active Treatment Arm; Crossover Active Treatment Arm
Device: Sham Acoustic Stimulation Therapy Device — The sham intervention uses the same device setup with sham procedures.
  Other Names: Sham SUI-100™ Device
  Arms: Sham Treatment Arm

SUMMARY:
The goal of this pivotal clinical trial is to evaluate the safety and effectiveness of the SUI-100 device for the treatment of mild-to-moderate stress urinary incontinence (SUI) in females aged 22-70 years.

The main questions this study aims to answer are:

1. Does treatment with the SUI-100 device reduce SUI symptoms, as measured by urine leakage.
2. Is the device safe and effective compared to the sham group?

Participants will:

1. Be randomly assigned to an active or sham control group in a blinded, multicenter study.
2. Attend treatment visits during the Treatment Phase, with SUI assessments conducted at specific intervals.
3. Enter a 3-month, treatment-free follow-up phase, with SUI assessment.
4. Proceed to three monthly maintenance treatments, followed by a final SUI assessment at study exit.

The total study duration will last approximately 18 months, with each individual's participation lasting approximately 6-8 months. This study aims to provide robust data on the effectiveness, safety, and durability of the SUI-100 device for treating female Stress Urinary Incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence, characterized by the involuntary loss of urine during activities that increase intra-abdominal pressure, affects approximately 50% of women with urinary incontinence and significantly impacts their quality of life. The SUI-100 device offers a novel, low-risk alternative to existing treatments, addressing a critical need for effective and conservative options.

Study Design:

The trial employs a randomized, blinded, sham-controlled, multi-center approach with an option for cross-over for participants randomized to sham.

Study Aim:

The study aims to determine the safety and efficacy of the study product in treating SUI. The study device is non-surgical and non-invasive.

Primary and Secondary Outcomes:

The study's primary objective is to determine whether treatment with the device reduces urine leakage by ≥50%, as measured by the 24-Hour Pad Weight Test, compared to the sham arm.

Safety Monitoring:

Safety assessments will be conducted throughout the study, with all adverse events (AEs) and adverse device effects (ADEs) documented and graded for severity.

Key Distinctions:

This trial is unique in its use of a non-invasive device that may offer a low-risk alternative to invasive treatments like urethral slings and radiofrequency therapy. The study's design, incorporating a sham-controlled, blinded methodology, ensures rigorous evaluation of the device's efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 22-70 years
2. MESA-UIQ SUI score must exceed MESA-UIQ UUI score
3. Investigator diagnosis of SUI at Baseline Study Visit A
4. µ-24-PWT >10 grams, and ≤74 grams
5. Positive PST (observed urine loss during coughing or Valsalva maneuver)
6. Able to independently read and willing to provide written informed consent and comply with all study visits and assessments required by study protocol
7. Able to independently read and complete all questionnaires and diaries provided in English
8. Negative urine test for urinary tract infection (UTI)
9. Negative urine test for pregnancy
10. Willing to use physician-approved contraception and avoid pregnancy for the duration of the study period if of child-bearing potential. An oral contraceptive may be started at study enrollment. Intrauterine device (IUD) is allowed if placed prior to study participation and not removed during the study.
11. Agrees not to participate in any other clinical research study(s) during this study
12. Willing to maintain same dose for any urge urinary incontinence (UUI) medications during study
13. If taking any of the following medications (may not start during trial); oral or vaginal estrogen therapy or other medication known to affect incontinence, such as testosterone, growth hormones, alpha-blockers, sedative-hypnotics, antipsychotics, angiotensin-converting enzyme (ACE) inhibitors, loop diuretics, and calcium channel blockers, must be stable for 3 months prior, and willing to maintain same dose throughout trial

Exclusion Criteria:

1. Body Mass Index (BMI) >35
2. µ-24-PWT ≥ 75 grams
3. Subject is non-ambulatory
4. Inability to maintain the low lithotomy position in a relaxed manner for the duration of the treatment delivery during visit
5. Subject has any electrical or electromagnetic implanted medical devices
6. History of UUI or mixed incontinence with a predominant urge component
7. History of incontinence of neurogenic etiology
8. Subject is pregnant or <12-months post-partum
9. Pelvic organ prolapse (POP) (e.g., greater than Stage 2 as defined by the International Continence Society (e.g., cystocele, rectocele)
10. PVR urine test volume >150 mL
11. Prior treatments for SUI:

    1. Any SUI surgery (e.g., slings)
    2. Bulking agent injection within 1 year
    3. Electrostimulation or magnetic stimulation within 3 months
    4. Pessary or urethral plug unless removed at least two weeks prior to start of study
    5. Physical therapy or pelvic floor exercises, such as Kegel exercises, to strengthen pelvic floor muscles and urinary sphincter within the past 60 days
12. Diagnosis of pelvic pain
13. History of radiation to the pelvis
14. Any recent pelvic surgery (within 1 year)
15. History of bladder stone
16. History of interstitial cystitis
17. History of dyspareunia or external vaginal pain syndromes such as vulvodynia
18. Hematuria
19. Neurological diseases known to affect the bladder
20. Conditions posing additional risks:

    1. Bleeding disorder or currently taking anticoagulants
    2. Current urinary infection - positive urine culture, signs of urinary infection; may repeat inclusion criteria urinary analysis (UA) after the UTI has been successfully resolved with a full course of antibiotics and a report UA is negative
    3. History of cervical, uterine, bladder, urethral, or rectal cancer
    4. Genital warts, lesions, or sexually transmitted disease that are locally visible
21. Currently undergoing any incontinence treatment
22. Concurrent enrollment in another clinical trial
23. Not suitable for the study or is at risk of study non-compliance in the judgement of the Principal Investigator (PI)

Ages: 22 Years to 77 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-11-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a ≥50% reduction in urine leakage. | Immediately following intervention.
  The proportion of participants achieving at least a 50% reduction in urine leakage as measured by the average of three 24-Hour Pad Weight Tests (µ-24-PWT).

SECONDARY OUTCOMES:
Percentage of participants with a ≥80% reduction in urine leakage. | Immediately following intervention.
  The proportion of participants achieving at least an 80% reduction in urine leakage as measured by the 24-Hour Pad Weight Test.
Percentage of participants with a ≥50% reduction in urine leakage after 10 treatments. | After 10 intervention treatments.
  The proportion of participants achieving at least a 50% reduction in urine leakage as measured by the average of three 24-Hour Pad Weight Tests (µ-24-PWT).
Percentage of participants maintaining a ≥50% reduction in urine leakage after the maintenance phase. | Immediately after treatments are complete for the study.
  The proportion of participants maintaining at least a 50% reduction in urine leakage after the maintenance phase.
Quality-of-life improvement using the Incontinence Impact Questionnaire-Short Form (IIQ-7). (Reduction in score means improvement min: 0, max 21) | Immediately following intervention.
  Reduction (improvement) in IIQ-7 scores by at least 30% from baseline.
Durability of treatment effects after the follow-up phase. | 3 months after intervention
  The proportion of participants maintaining a ≥50% reduction in urine leakage as measured by the average of three 24-Hour Pad Weight Tests (µ-24-PWT).

OTHER OUTCOMES:
Safety of the SUI-100 Device as determined by adverse events (AEs) and adverse device effects (ADEs). | Through study completion, an average of 9 months
  All AEs and ADEs will be monitored, documented, and graded for severity and relationship to the study device.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arizona Gynecology Consultants, Phoenix, Arizona
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Advanced Specialty Research, Boise, Idaho
  - Cypress Medical Research Center, Wichita, Kansas
  - Boeson Research GTF, Great Falls, Montana
  - Foundation for Female Health Awareness, Las Vegas, Nevada
  - Helios Clinical Research, Middleburg Heights, Ohio

IPD SHARING:
Plan to Share IPD: No